CLINICAL TRIAL: NCT07167160
Title: Camrelizumab Combined With Chemotherapy for Adjuvant Treatment of Cervical Cancer Patients With Pathologically Confirmed Lymph Node Positivity After Stage Surgery: A Prospective, Single-Arm, Multicenter, Phase II Clinical Trial
Brief Title: Chemo-immunotherapy for Cervical Cancer Stage IIICp Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20250023
Record Dates: First submitted 2025-09-01; First posted 2025-09-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer; Immunochemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy group (Experimental)
  Interventions: Drug: Camrelizumab combined with chemotherapy

INTERVENTIONS:
Drug: Camrelizumab combined with chemotherapy — Camrelizumab combined with chemotherapy for adjuvant treatment of patients with pathologically confirmed lymph node-positive cervical cancer after staging surgery

SUMMARY:
Efficacy evaluation of camrelizumab combined with chemotherapy for adjuvant treatment of patients with pathologically confirmed lymph node-positive cervical cancer after staging surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cervical cancer staged FIGO2018 IIIC1p or IIIC2p after radical surgery;
2. Positive PD-L1 expression;
3. ECOG score ≤1

Exclusion Criteria:

1. Positive parametrium or surgical margin;
2. Incomplete radical surgery;
3. Residual target lesions;
4. Active autoimmune disease or autoimmune disease requiring systemic treatment;
5. Previous treatment with immune checkpoint inhibitors.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate | from enrollment until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 100 months

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No